CLINICAL TRIAL: NCT05300503
Title: Evaluating the Use of a Remote Telehome Monitoring and Management Hypertension Program for Patients Receiving Virtual Care: A Pilot Randomized Controlled Trial
Brief Title: Evaluating the Use of a Remote Telehome Monitoring Hypertension Program for Patients Receiving Virtual Care
Acronym: HTMTHM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20210851-01H
Record Dates: First submitted 2022-03-18; First posted 2022-03-29 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-07

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in a 1:1 fashion to either the control group or intervention group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Participants will be asked to continue their usual day to day activities and take their current medications as directed. They will be sent a link by email or through MyChart to the standard video & education session on managing hypertension. They will watch the video at home on their own time. Participants will use a home blood pressure monitor to track their blood pressure (those without a blood pressure cuff will be provided one) for the 3-month intervention period. Patients will be provided instructions of when they should seek medical attention (clinical symptoms or SBP <100 or SBP >160). They will be encouraged to track their blood pressure daily and any symptoms they may be feeling.
- Intervention (Experimental): Participants will be asked to continue their usual day to day activities and take their current medications as directed. They will be sent a link by email or through MyChart to the educational session described above in the control group section. They will receive an Aetonix aTouchAway platform monitor, which is a disease specific home monitoring device to take home for 3 month intervention period. The device will prompt the participant to check their blood pressure on a daily basis and will send all readings to the UOHI Telehome monitoring program. The telehome monitoring nursing team will monitor the readings for each participant. For hypertensive patients who are not at target with their BP, the telehome monitoring nurse will titrate medications based on an advanced medical directive every 2 weeks. Patients will be provided instructions of when they should seek medical attention (clinical symptoms or SBP <100 or SBP >160).
  Interventions: Behavioral: Telehome Monitoring

INTERVENTIONS:
Behavioral: Telehome Monitoring — Participants are enrolled into the Telehome Monitoring program
  Arms: Intervention

SUMMARY:
High blood pressure or hypertension (HTN) is very common and can lead to serious health issues and even death. Medications and lifestyle changes can be used to treat HTN. During the Coronavirus Disease-19 (COVID-19) pandemic, a lot of the care provided by doctors has become virtual, meaning that patients can be assessed by a doctor over the phone or video call without needing to go to a clinic or hospital. Although this is convenient, a lot of people cannot get their blood pressure (BP) checked in a reliable way when they are at home. As a result, it is possible that their BPs are too high and that they are not getting the right medications or the right doses of medications to treat this. The Investigators are performing this study to see how patients are managing to check their BP's at home, during this time when a lot of the care is virtual. The Investigative team understands that many patients diagnosed with HTN don't have a home BP cuff, or might not know how to properly use it, or might not share the results with their doctors. In people who have high BP, we want to see if a special BP cuff and special monitoring program can help to get their BP's under better control, and to prevent negative effects related to HTN.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of primary, essential HTN (SBP>140/90mmHg or >130/80mmHg for diabetes)
* Have access to a phone (can be a landline)
* Have access to cellular (4G) network at their primary residence (they do not need to physically own a cellular phone but the need to be able to confirm their residence has 4G network access in order to connect the Aetonix aTouchAway platform to the network)
* Speak English or French

Exclusion Criteria:

* Patients who have been referred or who are actively managed at a specialized HTN clinic or other Telehome monitoring program
* Women who are pregnant, breastfeeding or planning to become pregnant
* Patients who are institutionalized at a retirement home, nursing home or long-term care facility
* Patients who plan on travelling out of the country for more than 2 weeks at any point during the intervention phase of the study (first 3 months)
* Patients who are cognitively impaired or experiencing acute psychiatric illness that would alter their ability to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-08-04 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Current state of blood pressure control in virtual settings | 3 months
  To document the status of blood pressure control (both systolic and diastolic) in virtual hypertension care settings.
Blood pressure response | 3 months
  Our primary outcome, which is the 24-hour ABPM, will be used to measure BP response in the control & intervention group at baseline & after 3-months of the intervention. We will repeat the 24-hour ABPM at 6-months follow up (3-months after completion of the intervention) to assess if there is maintenance of the intervention effects over time. Both systolic and diastolic measurements will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Mir, MD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (1):
- The University of Ottawa Heart Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
This this a pilot study, individual participant results will not be shared with other researchers.